CLINICAL TRIAL: NCT02003014
Title: Actos Tablets Special Drug Use Surveillance "Combined Use of Biguanides / Long-term Treatment"
Brief Title: Pioglitazone Tablets Special Drug Use Surveillance "Combined Use of Biguanides / Long-term Treatment"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 237-017; JapicCTI-132329 (Registry Identifier: JapicCTI); JapicCTI-R160828 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pioglitazone 15 mg to 30 mg: administered orally once daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone Tablets
  Other Names: Actos

SUMMARY:
To investigate the safety and efficacy of long-term treatment with pioglitazone (Actos tablets) in combination with biguanides (for 12 months after the start of pioglitazone tablets treatment) in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a special drug use surveillance with an observation period of 12 months designed to investigate the safety and efficacy of pioglitazone (Actos) in the routine clinical setting in patients with type 2 diabetes mellitus who responded inadequately to treatment with biguanides in addition to diet therapy and exercise therapy (planned sample size, 1000).

The usual adult dosage is 15 to 30 mg of pioglitazone administered orally once daily before or after breakfast. Dose adjustment will be made according to gender, age, and symptoms with an upper limit of 45 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus who responded inadequately to treatment with biguanides in addition to diet therapy and exercise therapy
2. Patients with available HbA1c data within the 1 month prior to the start of Actos Tablets treatment
3. Patients likely to be available for a 12-month observation after the start of Actos Tablets treatment

Exclusion Criteria:

1. Patients who have received Actos Tablets within the past 3 months.
2. Patients who started treatment with biguanides and Actos Tablets simultaneously
3. Patients who discontinued biguanides and switched to Actos Tablets treatment.
4. Patients who received additional biguanides after the start of Actos Tablets treatment
5. Patients with contraindications to Actos Tablets treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 152 investigative sites in Japan from 23 February 2009 to 31 January 2012.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who failed to respond adequately to treatment with biguanides were enrolled to receive pioglitazone 15 milligram (mg) - 30 mg for up to 12 months.
Groups:
- Pioglitazone: Pioglitazone 15 mg - 30 mg, tablet, orally, once daily for up to 12 months in participants based upon the disease severity.
Period: Overall Study
Arm/Group | Pioglitazone
Started | 899
Completed | 880
Not Completed | 19
Not completed — Case report forms uncollected | 9
Not completed — Treatment started after contract period | 1
Not completed — Patient did not visit the study site | 5
Not completed — Investigator's transfer | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Pioglitazone
Number analyzed (Participants) | 880
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 334
  Male | 546
Pregnancy status [Number; unit: participants] — The baseline characteristic was analyzed only in female participants.
  participants
    Not pregnant | 334
    Pregnant | 0
Time from diagnosis of type 2 diabetes [Number; unit: participants]
  Less than (<) 1 years | 36
  Greater than equal to (>=) 1 to <5 years | 194
  >=5 to <10 years | 239
  >=10 years | 354
  Unknown | 57
Predisposition to Hypersensitivity [Number; unit: participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  participants
    Had no predisposition to hypersensitivity | 856
    Had predisposition to hypersensitivity | 24
Details Regarding Predisposition to Hypersensitivity [Number; unit: participants] — Predisposition to hypersensitivity was categorized as hypersensitivity due to drug, food, or other. The baseline characteristic was analyzed in only participants who had a liability or tendency to suffer from hypersensitivity.
  participants
    Drug | 12
    Food | 5
    Other | 7
Drinking Habits [Number; unit: participants]
  None | 474
  Former drinker | 46
  Current drinker | 346
  Unknown | 14
Smoking Habits [Number; unit: participants]
  None | 520
  Former smoker | 145
  Current smoker | 203
  Unknown | 12
Weight [Number; unit: participants]
  < 40 kilogram (kg) | 3
  >=40 to <50 kg | 54
  >=50 to <60 kg | 163
  >=60 to <70 kg | 268
  >=70 kg | 384
  Unknown | 8
Body Mass Index [Number; unit: participants]
  < 18.5 kilogram per square meter (kg/m^2) | 14
  >=18.5 to <25 kg/m^2 | 382
  >=25 to <30 kg/m^2 | 346
  >=30 kg/m^2 | 124
  Unknown | 14
Medical History [Number; unit: participants]
  Had no presence of medical history | 672
  Had presence of medical history | 206
  Unknown | 2
Breakdown of Medical History [Number; unit: participants] — Breakdown of medical history was categorized as liver disease, renal disease, heart disease, cerebrovascular disease, malignant tumor and any other disease from those mentioned above. The baseline characteristic was analyzed only in participants who had medical history. Participants could be counted in more than 1 category (including duplicates).
  participants
    Liver disease | 6
    Renal disease | 4
    Heart disease | 20
    Cerebrovascular disease | 21
    Malignant tumor | 23
    Other | 154
Medical Complications [Number; unit: participants]
  Had no presence of medical complications | 100
  Had presence of medical complications | 780
Breakdown of Complications [Number; unit: participants] — Breakdown of medical complications was categorized as diabetic retinopathy,diabetic nephropathy,diabetic neuropathy,dyslipidaemia,hypertension,heart disease,liver disease(all types of liver disease),hepatic steatosis,alcoholic liver injury,viral liver injury,other liver disease,renal disease(other than diabetic nephropathy),renal disease(including diabetic nephropathy),malignant tumor,cerebrovascular disease,any other disease from those mentioned above.Baseline characteristic was analyzed only in participants who had medical complications. Participants could be counted in more than 1 category.
  participants
    Diabetic retinopathy | 63
    Diabetic nephropathy | 75
    Diabetic neuropathy | 58
    Dyslipidaemia | 217
    Hypertension | 203
    Heart disease | 85
    Liver disease (all types of liver disease) | 79
    Hepatic steatosis | 58
    Alcoholic liver injury | 11
    Viral liver injury | 1
    Other liver disease | 19
    Renal disease (other than diabetic nephropathy) | 14
    Renal disease (including diabetic nephropathy) | 85
    Malignant tumor | 8
    Cerebrovascular disease | 38
    Other | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 880
participants | 79

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAEs) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 880
participants | 1

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at 3 months, 6 months, 9 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline.
Time Frame: Baseline, Months 3, 6, 9, 12 and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Pioglitazone
Number analyzed (Participants) | 824
percentage of glycosylated hemoglobin
  Baseline (n = 824) | 8.34 (1.217)
  Change at Month 3 (n = 802) | -0.71 (0.943)
  Change at Month 6 (n = 721) | -0.79 (1.064)
  Change at Month 9 (n = 650) | -0.85 (1.066)
  Change at Month 12 (n = 624) | -0.91 (1.080)
  Change at Final Assessment (n = 824) | 0.85 (1.120)

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change between the fasting blood glucose value collected at 3 months, 6 months, 9 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline.
Time Frame: Baseline, Months 3, 6, 9, 12 and final assessment (up to Month 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Pioglitazone
Number analyzed (Participants) | 210
milligram per deciliter (mg/dL)
  Baseline (n = 210) | 174.1 (62.02)
  Change at Month 3 (n = 179) | -27.4 (59.41)
  Change at Month 6 (n = 152) | -27.9 (52.29)
  Change at Month 9 (n = 143) | -20.8 (65.77)
  Change at Month 12 (n = 146) | -28.4 (48.44)
  Change at Final Assessment (n = 210) | -28.1 (51.31)

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Change relative to baseline in participant's weight measured at 3 months, 6 months, 9 months, 12 months or final visit (last visit for a participant in the study, up to Month 12).
Time Frame: Baseline, Months 3, 6, 9, 12 and final assessment (up to Month 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 788
kg
  Baseline (n = 788) | 68.971 (14.1768)
  Change at Month 3 (n = 733) | 0.667 (1.9398)
  Change at Month 6 (n = 660) | 1.180 (2.4136)
  Change at Month 9 (n = 587) | 1.440 (2.6187)
  Change at Month 12 (n = 582) | 1.407 (2.7272)
  Change at Final Assessment (n = 788) | 1.465 (2.8322)

6. Secondary Outcome: Change From Baseline in Immunoreactive Insulin (IRI)
Description: The change in the value of IRI (portion of insulin in blood measured by immunochemical methods for the hormone; presumed to represent the free [unbound] and biologically active fraction of total blood insulin) collected at 3 months, 6 months, 9 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline.
Time Frame: Baseline, Months 3, 6, 9, 12 and final assessment (up to Month 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micro units per milliliter (mcU/mL)
Arm/Group | Pioglitazone
Number analyzed (Participants) | 44
micro units per milliliter (mcU/mL)
  Baseline (n = 44) | 10.320 (6.5620)
  Change at Month 3 (n = 29) | -1.390 (4.1813)
  Change at Month 6 (n = 32) | -2.438 (3.7622)
  Change at Month 9 (n = 20) | -2.970 (5.5698)
  Change at Month 12 (n = 27) | -1.774 (4.6780)
  Change at Final Assessment (n = 44) | -1.077 (4.7957)

7. Secondary Outcome: Change From Baseline Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: The change between homeostasis model assessment of insulin resistance collected at 3 months, 6 months, 9 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. Homeostasis Model assessment of insulin resistance Measures insulin resistance, calculated by insulin times glucose, divided by a constant (22.5). A higher score indicates higher insulin resistance.
Time Frame: Baseline, Months 3, 6, 9, 12 and final assessment (up to Month 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Pioglitazone
Number analyzed (Participants) | 43
HOMA-IR score
  Baseline (n = 43) | 3.92 (2.751)
  Change at Month 3 (n = 28) | -0.85 (2.173)
  Change at Month 6 (n = 31) | -1.41 (1.936)
  Change at Month 9 (n = 20) | -1.49 (2.779)
  Change at Month 12 (n = 26) | -1.26 (1.974)
  Change at Final Assessment (n = 43) | -0.75 (2.098)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in this study.
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 12/880
Other Adverse Events (participants affected / at risk) | 36/880
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=880)
Appendicitis (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Mania (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=880)
Oedema (General disorders) | 20
Weight Increased (Investigations) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.